CLINICAL TRIAL: NCT04611789
Title: A Randomized, Placebo-Controlled, Participant- and Investigator-Blind, Phase 1 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of LY3832479 Administered Subcutaneously to Healthy Participants
Brief Title: A Study of LY3832479 (LY-CoV016) in Healthy Participants 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18154; J2Z-MC-PGAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-10-30; First posted 2020-11-02 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — etesevimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3832479 (Experimental): Participants received single subcutaneous dose of 350 milligrams (mg) and 1000 mg LY3832479.
  Interventions: Drug: LY3832479
- Placebo (Placebo Comparator): Participants received single subcutaneous dose of Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3832479 — Administered subcutaneously
  Other Names: LY-CoV016; Etesevimab
  Arms: LY3832479
Drug: Placebo — Administered subcutaneously
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and tolerability of LY3832479 when it is given by injection just under the skin to healthy participants. Blood tests will be done to check how much LY3832479 is in the bloodstream and how long the body takes to eliminate it. Participation could last up to 16 weeks and may include up to six visits to the study center, with a one-week overnight stay.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history and physical examination
* Are willing to follow study procedures, including having nasal or nasopharyngeal swabs collected
* Have a body mass index (BMI) within the range of greater than or equal to (≥)18.5 to less than (<)35 kilograms per square meter (kg/m²)
* Male participants must agree to adhere to contraception restrictions
* Female participants must be of non-childbearing potential

Exclusion Criteria:

* Have or have had known or suspected severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection
* Have a history or presence of cardiovascular (including hypertension), respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disorders that, in the opinion of the investigator, are capable of

  * Significantly altering the absorption, metabolism, or elimination of drugs
  * Constituting a risk while taking the investigational product, or
  * Interfering with the interpretation of data
* Have significant allergies to humanized monoclonal antibodies (mAbs)
* Have any of the following that are clinically significant:

  * Multiple or severe drug allergies, or
  * Intolerance to topical corticosteroids, or
  * Severe posttreatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis)
* Have had lymphoma, leukemia, or any malignancy within the past 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Have had breast cancer within the past 10 years
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of current hepatitis C (that is, test positive for anti-hepatitis C antibody with confirmed presence of hepatitis C virus [HCV] ribonucleic acid [RNA])

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 350 mg LY3832479: Participants received single subcutaneous dose of 350 mg LY3832479.
- 1000 mg LY3832479: Participants received single subcutaneous dose of 1000 mg LY3832479.
Period: Overall Study
Arm/Group | Placebo | 350 mg LY3832479 | 1000 mg LY3832479
Started | 4 | 7 | 7
Completed | 3 | 7 | 7
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 350 mg LY3832479 | 1000 mg LY3832479 | Total
Number analyzed (Participants) | 4 | 7 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.8 (10.4) | 49.0 (12.4) | 42.7 (13.3) | 43.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 3 | 7
  Male | 4 | 3 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 4 | 9
  Not Hispanic or Latino | 1 | 5 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 4 | 4 | 6 | 14
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 7 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time 0 to Tlast (AUC[0-tlast]) of LY3832479
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Time 0 to tlast (AUC[0-tlast]) of LY3832479.
Time Frame: Day 1, 2, 3, 4, 5, 6, 7, 15, 29, 60 and 85 postdose
Population: All randomized participants who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (μg*day/mL)
Arm/Group | 350 mg LY3832479 | 1000 mg LY3832479
Number analyzed (Participants) | 7 | 7
microgram*day per milliliter (μg*day/mL) | 1560 (80) | 4530 (31)

2. Primary Outcome: PK: Maximum Serum Concentration (Cmax) of LY3832479
Description: PK: Maximum Serum Concentration (Cmax) of LY3832479.
Time Frame: Day 1, 2, 3, 4, 5, 6, 7, 15, 29, 60 and 85 postdose
Population: All randomized participants who received study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | 350 mg LY3832479 | 1000 mg LY3832479
Number analyzed (Participants) | 7 | 7
μg/mL | 39.1 (39) | 91.9 (35)

ADVERSE EVENTS:
Time Frame: Baseline, upto 3 Months
Description: All randomized participants.
Groups:
- Placebo SC: Participants received single subcutaneous dose of Placebo.
- 350 mg LY3832479 SC: Participants received single subcutaneous dose of 350 mg LY3832479.
- 1000 mg LY3832479 SC: Participants received single subcutaneous dose of 1000 mg LY3832479.
Arm/Group | Placebo SC | 350 mg LY3832479 SC | 1000 mg LY3832479 SC
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SC (N=4) | 350 mg LY3832479 SC (N=7) | 1000 mg LY3832479 SC (N=7)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT04611789/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT04611789/SAP_001.pdf